CLINICAL TRIAL: NCT03889886
Title: A Phase 2, Multicenter, Double-Masked, Randomized, Vehicle-Controlled, Parallel Group, Dose-Response Study of SDP-4 Ophthalmic Solution in Subjects With Dry Eye Disease (DED)
Brief Title: Study to Evaluate the Safety and Efficacy of SDP-4 in Subjects With Dry Eye Disease (DED)
Acronym: SDP-4-CS201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Silk Technologies, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SDP-4-CS201
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Results first posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2020-08

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to 1 of 3 concentrations (0.1%, 1.0% and 3.0%) of SDP-4 Ophthalmic Solution or vehicle in a 1:1:1:1 ratio in parallel groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All investigational product (SDP-4 concentrations and vehicle) will be provided in single-use doses (SUDs) contained in foil pouches.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Vehicle (Placebo Comparator): Vehicle
  Interventions: Drug: Vehicle
- SDP-4 Ophthalmic Solution (0.1%) (Experimental): Low concentration of SDP-4
  Interventions: Drug: SDP-4 Ophthalmic Solution (0.1%)
- SDP-4 Ophthalmic Solution (1.0%) (Experimental): Mid concentration of SDP-4
  Interventions: Drug: SDP-4 Ophthalmic Solution (1.0%)
- SDP-4 Ophthalmic Solution (3.0%) (Experimental): High concentration of SDP-4
  Interventions: Drug: SDP-4 Ophthalmic Solution (3.0%)

INTERVENTIONS:
Drug: SDP-4 Ophthalmic Solution (0.1%) — Investigational product (IP) will be administered via topical ocular instillation, one drop per eye, twice daily (BID) for 12 weeks (84 days). Both eyes will be treated.
  Other Names: SDP-4 (0.1%)
  Arms: SDP-4 Ophthalmic Solution (0.1%)
Drug: SDP-4 Ophthalmic Solution (1.0%) — Investigational product (IP) will be administered via topical ocular instillation, one drop per eye, twice daily (BID) for 12 weeks (84 days). Both eyes will be treated.
  Other Names: SDP-4 (1.0%)
  Arms: SDP-4 Ophthalmic Solution (1.0%)
Drug: SDP-4 Ophthalmic Solution (3.0%) — Investigational product (IP) will be administered via topical ocular instillation, one drop per eye, twice daily (BID) for 12 weeks (84 days). Both eyes will be treated.
  Other Names: SDP-4 (3.0%)
  Arms: SDP-4 Ophthalmic Solution (3.0%)
Drug: Vehicle — Investigational product (IP) will be administered via topical ocular instillation, one drop per eye, twice daily (BID) for 12 weeks (84 days). Both eyes will be treated.
  Arms: Vehicle

SUMMARY:
SDP-4-CS201, is a Phase 2, multi-center, double-masked, randomized, vehicle-controlled, dose-response, parallel-group study designed to evaluate the ocular and systemic safety and efficacy of SDP-4 ophthalmic solution in subjects with moderate to severe dry eye disease over a 12-week treatment period. Three concentrations (0.1%, 1.0% and 3.0%) of SDP-4 ophthalmic solution will be given to parallel groups via topical ocular instillation BID.

ELIGIBILITY:
Inclusion Criteria:

* Have DED in both eyes for ≥ 6 months prior to Visit 1/Screening.
* Total score ≥ 40 on the SANDE questionnaire.
* Tear break-up time (TBUT) of ≤ 6 seconds in both eyes.
* Anesthetized Schirmer's test tear volume ≥ 4 mm and <10 mm in both eyes.

Exclusion Criteria:

* Ocular surface corneal disease, other than DED.
* Lid margin disorder other than meibomian gland dysfunction (MGD).
* Any previous reconstructive or cosmetic eyelid surgery that may affect the normal function of the lids
* Any previous invasive glaucoma and/or corneal surgery
* Corneal refractive surgery in the 12 months prior to Visit 1/Screening.
* Cataract extraction within 90 days prior to Visit 1/Screening.
* Use of ophthlamic corticosteroids, NSAIDs, antibiotics, antihistamines, IOP lowering medication, in the 30 days prior to Visit 1/Screening
* Serious systemic disease or uncontrolled medical condition that in the judgment of the Investigator could confound study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Christensen, Study Director — Silk Technologies
Locations (26):
- United States (26):
  - Canyon City Eyecare, Azusa, California
  - Orange County Ophthalmology Medical Group, Garden Grove, California
  - North Valley Eye Medical Group, Mission Hills, California
  - LoBue Laser and Eye Medical Center, Murrieta, California
  - Eye Research Foundation, Newport Beach, California
  - North Bay Eye Associates, Petaluma, California
  - Grutzmacher & Lewis, A Medical Corporation DBA Sacramento Eye Consultants, Sacramento, California
  - Danbury Eye Physicians and Surgeons, PC, Danbury, Connecticut
  - Hernando Eye Institute, Brooksville, Florida
  - Eye Associates of Fort Myers, Fort Myers, Florida
  - Shettle Eye Research, Largo, Florida
  - West Coast Eye Institute, Lecanto, Florida
  - Clayton Eye Clinical Research, LLC, Morrow, Georgia
  - Coastal Research Associates, Roswell, Georgia
  - Kannarr Eye Care, Pittsburg, Kansas
  - Heart of America Eye Care, P.A., Shawnee Mission, Kansas
  - Ophthalmology Associates, St Louis, Missouri
  - Comprehensive Eye Care Ltd, Washington, Missouri
  - Wake Forest Health Network Ophthalmology- Oak Hollow, High Point, North Carolina
  - Drs. Quinn, Foster & Associates, Athens, Ohio
  - Abrams Eye Center, Cleveland, Ohio
  - Total Eye Care, Memphis, Tennessee
  - Eye Specialty Group, Memphis, Tennessee
  - Nashville Vision Associates, Nashville, Tennessee
  - Texan Eye / Keystone Research, Ltd., Austin, Texas
  - Medical Center Ophth Assoc / Keystone Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (0.1%) | SDP-4 Ophthalmic Solution (1.0%) | SDP-4 Ophthalmic Solution (3.0%)
Started | 76 | 77 | 76 | 76
Completed | 76 | 76 | 75 | 69
Not Completed | 0 | 1 | 1 | 7
Not completed — Other | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (0.1%) | SDP-4 Ophthalmic Solution (1.0%) | SDP-4 Ophthalmic Solution (3.0%) | Total
Number analyzed (Participants) | 76 | 77 | 76 | 76 | 305
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (15.2) | 60.5 (15.86) | 60.1 (15.58) | 61.5 (13.68) | 60.3 (15.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 64 | 61 | 64 | 245
  Male | 20 | 13 | 15 | 12 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 12 | 11 | 42
  Not Hispanic or Latino | 66 | 68 | 64 | 65 | 263
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 4 | 1 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 10 | 7 | 8 | 14 | 39
  White | 64 | 66 | 66 | 61 | 257
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Symptom Assessment in Dry Eye (SANDE) Questionnaire
Description: Mean change from baseline in total SANDE score at Visit 7/Day 84
  The SANDE questionnaire contained two questions regarding the frequency and severity of DED symptoms, with a total score being the square root of the frequency score times the square root of the severity score (range 0 100). A higher score indicates more severe DED symptoms.
Time Frame: 84 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (0.1%) | SDP-4 Ophthalmic Solution (1.0%) | SDP-4 Ophthalmic Solution (3.0%)
Number analyzed (Participants) | 76 | 76 | 75 | 69
units on a scale | -25.66 (26.685) | -25.14 (25.076) | -29.95 (24.883) | -24.81 (26.685)

2. Secondary Outcome: Tear Breakup Time
Description: Mean change from baseline at each visit
Time Frame: 84 days
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (0.1%) | SDP-4 Ophthalmic Solution (1.0%) | SDP-4 Ophthalmic Solution (3.0%)
Number analyzed (Participants) | 76 | 76 | 75 | 69
seconds
  Day 7 | 0.95 (1.816) | 1.29 (4.433) | 1.21 (2.993) | 0.80 (3.085)
  Day 14 | 1.08 (3.430) | 1.15 (1.487) | 1.37 (2.735) | 1.09 (2.175)
  Day 28 | 1.00 (2.246) | 1.92 (4.135) | 2.20 (4.498) | 1.63 (3.750)
  Day 56 | 1.18 (2.728) | 1.38 (2.020) | 2.13 (4.123) | 1.29 (1.878)
  Day 84 | 1.44 (3.213) | 1.44 (2.097) | 1.49 (3.177) | 1.09 (1.693)

3. Secondary Outcome: Anesthetized Schirmer's Test
Description: Mean change from baseline at Visit7/Day 84
Time Frame: 84 days
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (0.1%) | SDP-4 Ophthalmic Solution (1.0%) | SDP-4 Ophthalmic Solution (3.0%)
Number analyzed (Participants) | 76 | 76 | 75 | 69
millimeter | 2.53 (5.582) | 2.95 (6.190) | 1.89 (4.706) | 3.75 (5.699)

4. Secondary Outcome: Conjunctival Hyperemia
Description: Mean change from baseline at each visit.
  Reported on a scale of 0-15 with values greater than 3 indicating abnormal incidence of conjunctival surface irregularity.
Time Frame: 84 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (0.1%) | SDP-4 Ophthalmic Solution (1.0%) | SDP-4 Ophthalmic Solution (3.0%)
Number analyzed (Participants) | 76 | 76 | 75 | 69
units on a scale
  Day 7 | -0.6 (1.87) | -0.7 (1.82) | -0.9 (1.91) | -0.6 (2.19)
  Day 14 | -0.6 (2.28) | -0.8 (1.78) | -0.6 (2.28) | -0.6 (1.97)
  Day 28 | -0.8 (2.70) | -0.8 (1.98) | -0.9 (2.14) | -0.6 (2.59)
  Day 56 | -0.9 (2.30) | -0.6 (1.99) | -0.7 (2.48) | -0.7 (2.55)
  Day 84 | -0.6 (2.35) | -0.8 (2.60) | -0.3 (2.45) | -0.6 (2.16)

5. Secondary Outcome: Corneal Fluoroscein Staining
Description: Mean change from baseline at each visit
  Reported on a scale of 0-15 with values greater than 3 indicating abnormal incidence of corneal surface irregularity.
Time Frame: 84 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (0.1%) | SDP-4 Ophthalmic Solution (1.0%) | SDP-4 Ophthalmic Solution (3.0%)
Number analyzed (Participants) | 76 | 76 | 75 | 69
units on a scale
  Day 7 | -0.2 (2.15) | -1.4 (2.03) | -0.9 (2.16) | -1.4 (2.00)
  Day 14 | -0.5 (2.02) | -1.2 (2.21) | -1.1 (1.99) | -1.3 (2.11)
  Day 28 | -0.9 (2.55) | -1.5 (2.43) | -1.3 (1.97) | -1.2 (2.15)
  Day 56 | -1.2 (2.36) | -1.3 (2.07) | -0.9 (2.53) | -1.6 (1.96)
  Day 84 | -0.8 (1.96) | -1.3 (2.45) | -1.2 (2.99) | -1.4 (2.29)

ADVERSE EVENTS:
Time Frame: 84 days
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (0.1%) | SDP-4 Ophthalmic Solution (1.0%) | SDP-4 Ophthalmic Solution (3.0%)
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/76 | 0/75 | 0/69
Serious Adverse Events (participants affected / at risk) | 1/76 | 0/76 | 0/75 | 0/69
Other Adverse Events (participants affected / at risk) | 15/76 | 14/76 | 16/75 | 23/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=76) | SDP-4 Ophthalmic Solution (0.1%) (N=76) | SDP-4 Ophthalmic Solution (1.0%) (N=75) | SDP-4 Ophthalmic Solution (3.0%) (N=69)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — One subject was hospitalized for diverticulitis and recovered. The event was judged not related to treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=76) | SDP-4 Ophthalmic Solution (0.1%) (N=76) | SDP-4 Ophthalmic Solution (1.0%) (N=75) | SDP-4 Ophthalmic Solution (3.0%) (N=69)
Eye Disorders (Eye disorders) | 8 (11) | 9 (13) | 9 (12) | 16 (28) — Category containing a number of different, minor eye conditions.
General Disorders and administration site conditions (General disorders) | 6 (6) | 5 (5) | 10 (10) | 6 (7) — Installation site pain
Investigations (Investigations) | 2 (2) | 1 (2) | 0 (0) | 1 (1) — Intraocular pressure increased Vital dye staining cornea present

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information concerning SDP-4 and the operations of Silk Technologies, such as patent applications, formulas, manufacturing processes, basic scientific data or formulation information not previously published, are considered CONFIDENTIAL and shall remain the sole property of Silk Technologies. The Investigator agrees to use this information only in accomplishing this study and will not use it for other purposes without the written consent of Silk Technologies

DOCUMENTS (3):
  • Study Protocol (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT03889886/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/86/NCT03889886/SAP_001.pdf
  • Informed Consent Form (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/86/NCT03889886/ICF_002.pdf